CLINICAL TRIAL: NCT03327870
Title: Oral Health Needs Assessment of Sjogren's Syndrome and Salivary Gland Dysfunction Cohorts and Healthy Volunteers - Evaluating Oral Health Disparities as Determinants of Oral Health in a High-risk Population
Brief Title: Oral Health Needs Assessment of Sjogren s Syndrome and Salivary Gland Dysfunction Cohorts and Healthy Volunteers Evaluating Oral Health Disparities as Determinants of Oral Health in a High-Risk Population
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180007; 18-D-0007
Record Dates: First submitted 2017-10-31; First posted 2017-11-01 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Sjogren's Syndrome; Oral Health
Keywords: Sjogren's Syndrome; Sicca
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (5):
- 1: Sjogren's Syndrome
- 2: Sicca
- 3: Incomplete Sjogren's Syndrome
- 4: Healthy Volunteers
- 5: Excluded by 2016 ACR/EULAR Classificastion Criteria

SUMMARY:
Background:

A person s dental health depends on many factors. Some are social, economic, or behavioral. Some are environmental. People with Sj(SqrRoot)(Delta)gren s Syndrome have a change in the amount and quality of saliva. This may affect dental health. Researchers want to study the dental health needs of people with this and other salivary gland problems. They will compare these findings with healthy volunteers. This will help them improve health care for these groups of people.

Objectives:

To study dental health needs of people with salivary gland problems and healthy volunteers. To study the disparities in dental health between these groups.

Eligibility:

Adults 18 and older who were in a Sj(SqrRoot)(Delta)gren s Syndrome study

Healthy volunteers the same age

Design:

Participants will take an online survey. It should take less than 30 minutes. They can skip any questions.

They will be asked about dental health, general health, and well-being.

Information in the survey will be kept secure.

DETAILED DESCRIPTION:
Objective:

Determinants of health, particularly oral health, have not been evaluated in the context of Sjogren s Syndrome (SS) and other salivary gland dysfunctions. It is known that the quantitative and qualitative changes in salivary flow that occur in SS place those with this complex autoimmune disorder at increased risk of dental caries, oral infections, mucosal ulceration, salivary gland enlargement and functional impairment. There is conflicting evidence on the risk of periodontal disease in this population. Furthermore, it has been reported that this population experiences a greater number of dental visits, decayed teeth, and dental restorations in the preceding year, and have a 2-3 fold increased annual out-of pocket dental care expenditure compared to those without SS. Moreover, the oral and dental needs of those with SS have not been quantified in the context of oral health disparities, i.e., by strata of vulnerable groups. Those with other salivary gland dysfunction such as Sicca and those who have signs and symptoms of salivary gland dysfunction that only partially fulfill the classification criteria for SS, also known as incomplete SS (ISS), have neither been assessed for oral health needs nor have oral health disparities been ascertained in this high-risk population.

Study Population:

We will enroll adults classified as SS, Sicca, ISS, as well healthy volunteers as well as those excluded by the 2016 ACR/EULAR classification criteria for SS. Therefore, the aims of this study are to:

1. Ascertain the oral health needs of those with SS, Sicca, and ISS in comparison with healthy volunteers (HV)
2. Identify oral health disparities in this high-risk population (SS, Sicca, ISS) in comparison with HV.

Design:

This will be an observational study with a cross-sectional survey administered to the study population at enrollment, to ascertain their oral health needs and oral health disparities.

Outcome Measures:

Study participants have been evaluated and classified into SS, Sicca, ISS, and HV cohorts as part of the SS clinical protocols: 84-D-0056, 99-D-0018, 11-D-0172, 15-D-0051 and 94-D-0018.

A. Primary outcome

Oral Health Outcomes will be captured using the protocols described in the NHANES Oral Health Questionnaire, with the inclusion of additional dental/oral health questions. All oral health outcomes will be ascertained once at the time of study enrollment. Self-reported oral health needs and self-reported importance of key oral health needs will be ascertained as part of the double-scaled oral health study instrument. This will enable discrepancy scoring of key oral health outcomes and calculation of a numeric needs index. These instruments have been pilot tested.

B. Exposures

Oral Health Disparities will be based on indicators for the following and will be ascertained at enrollment:

* Age
* Race
* Ethnicity
* SES levels (Educational attainment, employment status, home ownership, food security)
* Geographic location (Six-level urban-rural classification scheme for U.S. counties and county-equivalent entities developed by NCHS).
* Gender
* Sexual orientation
* Marital status
* Disabilities (physical disability)
* Mental health

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects enrolled in 94-D-0018, 11-D-0172, 15-D-0051 and previously enrolled in 84-D-0056 and 99-D-0070

EXCLUSION CRITIERIA:

* NIH employees working at NIDCR and under the supervision of SSGDU supervisors.
* Those less than 18 years of age.
* Those unable to give consent
* Those unable to speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults classified as Sjogren's Syndrome (SS), Sicca, ISS, as well healthy volunteers as well as those excluded by the 2016 ACR/EULAR classification criteria for SS.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Self-reported oral health needs and importance of key oral health indicators are the outcomes | Survey completion

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Iafolla, D.M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States